CLINICAL TRIAL: NCT06712823
Title: An Open-label, Long-term Extension Study to Evaluate Safety and Efficacy in Participants Treated With CRN04894
Brief Title: An Extension Study to Evaluate Safety and Efficacy in Participants Treated With CRN04894
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Crinetics Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRN04894-09; 2024-514846-35-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-27; First posted 2024-12-02 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-06

CONDITIONS: Congenital Adrenal Hyperplasia; Classic Congenital Adrenal Hyperplasia
Keywords: Congenital Adrenal Hyperplasia; CAH; CRN04894; atumelnant
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Open-label treatment period (up to 2 years). The maximum atumelnant dose permitted is not to exceed the highest atumelnant dose explored in a parent study for the indication.
  Interventions: Drug: atumelnant (CRN04894)

INTERVENTIONS:
Drug: atumelnant (CRN04894) — Atumelnant is an orally active nonpeptide melanocortin 2 receptor (MC2R) or adrenocorticotropic hormone (ACTH) receptor antagonist.

SUMMARY:
The purpose of this study is to evaluate the long-term safety, tolerability, and efficacy of atumelnant (CRN04894).

DETAILED DESCRIPTION:
This single-arm, long-term, open-label, study is designed to evaluate the safety, tolerability, and efficacy of atumelnant (CRN04894) in participants with congenital adrenal hyperplasia (CAH). Enrollment will be limited to individuals who completed a parent study with CRN04894 or completed treatment in a Crinetics atumelnant study, and in the opinion of the Investigator had an acceptable benefit-risk assessment in the completed study and would benefit from continued dosing in this extension study.

Approximately 150 participants will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all the following criteria apply:

1. Participants with CAH who have completed a Crinetics CRN04894 study or completed treatment in a Crinetics CRN04894 study, and in the opinion of the Investigator had an acceptable benefit-risk assessment in the completed study and would benefit from continued dosing in this extension study.
2. Participants must be compliant, in the opinion of the Investigator, with a stable regimen of glucocorticoid replacement (eg, hydrocortisone, prednisolone, prednisone, methylprednisolone), and be taking a daily dose of hydrocortisone (HC) or equivalent at the time of Informed Consent.
3. Female participants who engage in heterosexual intercourse must:

   1. Be of nonchildbearing potential, defined as either surgically sterile (ie, hysterectomy, bilateral salpingectomy, tubal ligation for at least 3 months, or bilateral oophorectomy), OR
   2. Be postmenopausal with at least 1 year of amenorrhea. In participants with less than 1 year of amenorrhea, confirmation is required with 2 follicle-stimulating hormone (FSH) measurements. A documented, historical test result measured prior to Screening may be used as 1 of the 2 measurements. The FSH value should be ≥30 IU/L to confirm menopausal status, OR
   3. Agree to use a highly effective method of contraception from the beginning of Screening until at least 2 weeks after the last dose of study drug. Contraceptive use by men and women also should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. Periodic abstinence (ie, calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception.
4. Male participants agree to use a condom when sexually active with a female partner of childbearing potential from Screening until at least 2 weeks after the last dose of study drug (or be surgically sterile [ie, vasectomy with a confirmed absence of sperm in ejaculate]; or agree to remain abstinent on a long-term and persistent basis). Male participants should also agree to not donate sperm for the duration of the study and until at least 2 weeks after the last dose of study drug.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Any medical condition(s) or laboratory findings that, in the opinion of the Investigator, might jeopardize the participant's safety or ability to complete the study.
2. Participants have known history of (that is within the past 12 months), or current alcohol or drug abuse.
3. Participants have any mental condition rendering him/her unable to understand the nature, scope, and possible consequences of the study, and/or evidence of poor compliance with medical instructions.
4. Participants have a known allergy or hypersensitivity to any of the test materials or related compounds, including being at high risk of adrenal insufficiency as judged by the Investigator.
5. Women who are pregnant or lactating or, if of childbearing potential, who are unwilling to use highly effective contraception as described in this study. Male participants who are unwilling to use highly effective contraception as described in this study.
6. Participant is an employee or immediate family member of an employee of Crinetics.
7. Participants who have been dosed with an investigational drug (other than atumelnant) in any prior clinical study within 60 days or 5 half-lives (whichever is longer) prior to informed consent or plan to use an investigational drug in another study.
8. Participants with a history of cancer excluding cured/treated dermal squamous or basal cell carcinoma or cervical carcinoma in situ.
9. Participants who are committed to an institution by virtue of an order issued either by the judicial or the administrative authorities.

   Specific for Participants Not Currently Receiving Atumelnant
10. Participants with any clinically significant abnormal laboratory test during Screening or clinically significant concomitant disease other than CAH including but not limited to cardiovascular disease; moderate or severe renal insufficiency (estimated glomerular filtration rate <60 mL/min/1.73 m2 using Chronic Kidney Epidemiology Collaboration [CKD-EPI] formula) at Screening; or Significant liver disease or alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >3× upper limit of normal (ULN), and/or total bilirubin >1.5×ULN during Screening. Participants with previously diagnosed Gilbert's syndrome not accompanied by other hepatobiliary disorders and associated with total bilirubin <3.5 mg/dL (<51.3 μmol/L) will be permitted.
11. Participants with a history of bilateral adrenalectomy, hypopituitarism, or other condition requiring chronic glucocorticoid therapy.
12. Participants with a history of major surgery/surgical therapy for any cause within 4 weeks prior to Screening.
13. Participants with poorly controlled diabetes mellitus defined as having a hemoglobin A1c (HbA1c) ≥8.5% (≥69 mmol/mL).
14. Participants with hypothyroidism who are not receiving adequate hormone replacement therapy based on thyroid hormone levels measured at the time of Screening, as determined by the Investigator.
15. Participant has an average (of 3 electrocardiograms [ECGs]) Fridericia's corrected QT (QTcF) interval >450 milliseconds (msec) (men) or >470 msec (women), time interval between P and R waves (PR interval) >220 msec, time interval of the QRS complex (QRS) interval >120 msec, second- or third-degree atrioventricular block, left bundle branch block, or hemiblock at Screening.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) leading to discontinuation | Week 108
Incidence of glucocorticoid (GC) deficiency / adrenal insufficiency and adrenal crisis | Week 108
Incidence of hospitalizations related to congenital adrenal hyperplasia (CAH) | Week 108
Change from baseline in morning (before 11:00 AM) serum androstenedione (A4) over time | Week 108

SECONDARY OUTCOMES:
Change from baseline in morning (before 11:00 AM) serum 17-hydroxyprogesterone (17-OHP) over time | Week 108
Change from baseline in daily glucocorticoid (GC) dose (hydrocortisone [HC] mg equivalents) over time | Week 108

CONTACTS AND LOCATIONS:
Locations (9):
- United States (2):
  - Crinetics Study Site, Minneapolis, Minnesota 55454, Minneapolis, Minnesota
  - Crinetics Study Site, Morehead City, North Carolina
- Crinetics Study Site, Córdoba, Córdoba Province, Argentina
- Brazil (2):
  - Crinetics Study Site, Botucatu, São Paulo
  - Crinetics Study Site, São Paulo
- Crinetics Study Site, Munich, Bavaria, Germany
- Crinetics Study Site, Roma, Italy
- United Kingdom (2):
  - Crinetics Study Site, Birmingham
  - Crinetics Study Site, London

IPD SHARING:
Plan to Share IPD: No